CLINICAL TRIAL: NCT02956577
Title: Systolic and Diastolic Left Ventricular Function in Patients With Type 2 DIABetes Mellitus: Changes Over Time and Comparison With Cardiac Microcirculation. An ECHOcardiographic Study
Brief Title: Cardiac Function and Microcirculation: Type 2 DIABetes and ECHOcardiographic Changes Over Time
Acronym: DIABECHO
Status: Completed | Type: Observational
Sponsor: Svendborg Hospital (Other)
Responsible Party: Principal Investigator, Gokulan Pararajasingam, MD, Ph.D-student, Svendborg Hospital
Other Study IDs: OUHSVB001
Record Dates: First submitted 2016-10-30; First posted 2016-11-07 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Left Ventricular Dysfunction
Keywords: Global Longitudinal Strain (GLS); Coronary Flow Velocity Reserve (CFVR); Cardiac dysfunction; Microcirculation; Coronary Computed Tomography Angiography (CCTA); Type 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Ventricular Dysfunction, Left; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Storage in biobank (-80° C):
  5 x 2 ml (serum).
  4 x 2 ml (ethylenediaminetetraacetic acid).
  2 x 2 ml (sodium citrate)
  1 x 2 ml (erythrocyte sedimentation rate)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- T2: Patients with type 2 diabetes without myocardial infarction, heart failure and symptoms of cardiac disease at inclusion, were invited from the Outpatient Clinic of Endocrinology or The Eye Photo Clinic at Odense University Hospital (OUH) Svendborg. Diagnosis of diabetes was classified by trained endocrinologists according to international standards with relevant biochemistry. Historical data on urine- and blood samples as well as micro- and macrovascular diabetic complications have been registered consecutively in patients followed at the outpatient clinic in the regional Funen Diabetes Database (FDDB). Data on historical invasive procedures due to cardiac disease were registered in Western Denmark Heart Registry (WDHR).
- T1: Patients with type 1 diabetes without myocardial infarction, heart failure and symptoms of cardiac disease at inclusion, were invited from the Outpatient Clinic of Endocrinology or The Eye Photo Clinic at OUH Svendborg. Diagnosis of diabetes was classified by trained endocrinologists according to international standards with relevant biochemistry. Historical data on urine- and blood samples as well as micro- and macrovascular diabetic complications have been registered consecutively in patients followed at the outpatient clinic in the regional FDDB. Data on historical invasive procedures due to cardiac disease were registered in WDHR.
- Non-diabetic subjects: Non-diabetic subjects without myocardial infarction, heart failure and symptoms of cardiac disease at inclusion, were included from The Danish Cardiovascular Screening trial (DANCAVAS). A randomized controlled trial with the primary aim to evaluate the health benefits and costeffectiveness of using non-contrast full truncus computer tomography (CT) scans (to measure coronary artery calcification (CAC) and identify aortic/iliac aneurysms) and measurements of the ankle brachial blood pressure index (ABI) as part of a multifocal screening and intervention program for cardiovascular disease in men aged 65-74.

SUMMARY:
The purpose of this study was to investigate the influence of micro- and macrovascular changes on the cardiac function in relation to left ventricular function and coronary arteries during one year in patients with type 2 diabetes.

DETAILED DESCRIPTION:
The most frequent heart disease in patients with Type 2 Diabetes Mellitus (T2DM) is the premature development of coronary atherosclerosis, which often leads to overt ischemic heart disease (IHD). T2DM can lead to both cardiac dysfunction due to IHD or to diabetic cardiomyopathy. Diabetic cardiomyopathy is defined as an impairment of left ventricular (LV) function without overt obstructive coronary vessel disease. Diabetic cardiomyopathy has been associated with microvascular dysfunction, which leads to the inability of the heart to circulate blood effectively. The microvascular atherosclerotic changes are well known in patients with diabetes, such as impaired vision, kidney function and sensibility. The macrovascular atherosclerotic changes such as plaques in the coronary arteries are strongly associated with reduced left ventricular function.

However, the relationship between micro- and macrovascular atherosclerotic changes and the impact on cardiac function is less certain.

Estimation of cardiac function includes: Left Atrial (LA) Strain, LA Strain Rate (SR), LA Emptying Function (LAEF), LV Ejection Fraction (EF), Fractional Shortening (FS), Global Longitudinal Strain (GLS), Circumferential Strain (CS) and Radial Strain (RS), Strain Rate (SR), Peak Systolic Strain, Post Systolic Strain, Early mitral filling velocity (E), late mitral filling velocity (A), E/A ratio, Deceleration Time (DCT) of early mitral filling velocity, medial and lateral mitral velocities using tissue doppler (e' , a' and s'), E/e' ratio, Isovolumetric Relaxation Time (IVRT), Isovolumetric Closing Time (IVCT), Ejection Time (ET), Myocardial Performance Index (MPI) and Myocardial Work Index (MWI).

In this study, participants will be consisting of non-diabetic subjects and patients with diabetes type 1 + 2. All of the participants have no history of myocardial infarction, heart failure and current symptoms of cardiac disease.

The study population will undergo following examinations:

1. 12-lead electrocardiogram (ECG)
2. Urine- and blood samples.
3. Measurements of anthropometric data and vital parameters
4. Recording of medical history
5. 2D transthoracic echocardiography
6. Coronary flow velocity reserve (CFVR) with adenosine infusion.
7. Coronary computed tomography angiography (CCTA).
8. Free fractional reserve computed tomography (FFR-CT)

The examinations will be repeated at follow-up (however non-diabetic subjects will only have 1 CCTA performed at baseline).

The non-invasive FFR-CT will only be performed once in a subgroup of diabetic patients and non-diabetic subjects from November 2016 until May 2017.

ELIGIBILITY:
Inclusion criteria:

* Ability to give informed consent
* Estimated glomerular filtration rate (eGFR) > 45 ml/min
* NYHA I + II

Exclusion criteria:

* 2° or 3° AV-block at baseline
* Long QT-syndrome at baseline
* Sinus node dysfunction with long sinus arrest at baseline
* Angina pectoris at baseline
* Ejection fraction (EF) < 40% at baseline
* Atrial fibrillation at baseline
* Usage of dipyridamol at baseline
* Aortic stenosis and left ventricle hypertrophia at baseline
* Aortic insufficiency and left ventricle dilatation at baseline
* Medication for asthma within the last 4 years prior to baseline
* Medication for chronic obstructive pulmonary disease (COPD) at baseline
* Allergy to contrast agent at baseline
* Significant stenosis in left main (LM) / left anterior descending (LAD) artery at baseline
* Not feasible to measure or perform coronary flow velocity reserve (CFVR)
* Poor quality of echocardiographic images
* History of pacemaker
* History of myocardial infarction (MI)
* History of heart failure (HF)
* History of coronary artery bypass grafting (CABG)
* History of aortic valve replacement
* History of atrial fibrillation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetes type 1+2 and non-diabetic subjects from the DANCAVAS trial (NCT00662480)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Changes in Global Longitudinal Strain (GLS) stratified by Coronary Artery Calcium Score (CAC) in patients with diabetes during one year of follow-up | baseline, 12 months
  To evaluate the changes in GLS stratified by CAC during one year of follow-up in patients with diabetes compared to non-diabetic subjects

SECONDARY OUTCOMES:
Changes in GLS stratified by Coronary Flow Velocity Reserve (CFVR) in patients with diabetes during one year of follow-up | baseline, 12 months
  To evaluate the changes in GLS stratified by CFVR during one year of follow-up in patients with diabetes compared to non-diabetic subjects
Correlation between biomarkers and GLS stratified by CFVR | 12 months
  To evaluate the correlation between biomarkers (C-Reactive Protein, Troponin T, NT-proBNP and Uric Acid) and GLS stratified by CFVR in diabetic patients compared to non-diabetic subjects
Correlation between biomarkers and GLS stratified by CAC | 12 months
  To evaluate the correlation between biomarkers (C-Reactive Protein, Troponin T, NT-proBNP and Uric Acid) and GLS stratified by CAC in diabetic patients compared to non-diabetic subjects
Changes in LV function stratified by CAC | baseline, 12 months
  To evaluate LV systolic and diastolic function stratified by CAC in patients with diabetes compared to non-diabetic subjects.
Changes in LV function stratified by CFVR | baseline, 12 months
  To evaluate LV systolic and diastolic function stratified by CFVR in patients with diabetes compared to non-diabetic subjects.
Changes in LV function stratified by micro- and macrovascular diabetic status | baseline, 12 months
  To evaluate changes in LV systolic and diastolic function in relation to albuminuria, retinopathy, neuropathy, diabetes duration and CAC.
Correlation between CFVR and Free Fractional Reserve -Computed Tomography (FFR-CT) | baseline
  To evaluate the correlation between CFVR and FFR-CT in a subgroup consisting of diabetic patients and non-diabetic subjects.
Correlation between GLS and FFR-CT | baseline
  To evaluate the correlation between GLS and non-invasive FFR-CT in a subgroup consisting of diabetic patients and non-diabetic subjects.
Changes in GLS in patients with long-term diabetes and no macrovascular disease | baseline
  To evaluate the impact of historical varying levels of HbA1c and cholesterols on GLS at baseline in patients with diabetes and no macrovascular disease.

OTHER OUTCOMES:
Relationship between strain values and framerate | baseline, 12 months
  To evaluate the changes in strain values dependant of framerate
Relationship between strain values and omitted myocardial segments | baseline, 12 months
  To evaluate the changes in strain values dependant of number of myocardial segments omitted
Correlation between dysglycaemia and Left Ventricle Mass (LVM) | Baseline
  To evaluate the impact of dysglycaemia on LVM in non-diabetic subjects compared to diabetic patients.
Left Ventricle (LV) and Left Atrial (LA) function stratified by New York Heart Association (NYHA) functional class | baseline
  To evaluate LV and LA systolic and diastolic function in relation to NYHA classification
Changes in cardiac systolic and diastolic function stratified by CAC during five years of follow-up in patients with diabetes | baseline, 60months
  To evaluate the changes in cardiac systolic and diastolic function stratified by CAC during five years of follow-up in patients with diabetes compared to non-diabetic subjects.
Changes in cardiac systolic and diastolic function stratified by CFVR during five years of follow-up in patients with diabetes | baseline, 60months
  To evaluate the changes in cardiac systolic and diastolic function stratified by CFVR during five years of follow-up in patients with diabetes compared to non-diabetic subjects.
Changes in cardiac systolic and diastolic function stratified by plaque morphology during five years of follow-up in patients with diabetes | baseline, 60months
  To evaluate the changes in cardiac systolic and diastolic function stratified by plaque morphology during five years of follow-up in patients with diabetes compared to non-diabetic subjects.
LA function stratified by CFVR | baseline
  To evaluate atrial function stratified by CFVR in patients with diabetes compared to non-diabetic subjects.
LA function stratified by micro- and macrovascular status | baseline
  To evaluate atrial function in relation to albuminuria, retinopathy, neuropathy, diabetes duration and CAC.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Egstrup, DMSci, Study Director — Odense University Hospital (OUH) Svendborg Hospital
Locations (1):
- Cardiovascular Research Unit, OUH Svendborg Hospital, Svendborg, Denmark

IPD SHARING:
Plan to Share IPD: No